CLINICAL TRIAL: NCT07254156
Title: A Prospective, Multicenter, Exploratory Clinical Study Evaluating the Application of Tissue-Agnostic Technology in the Dynamic Monitoring of Minimal Residual Disease in Stage III Colorectal Cancer
Brief Title: A Study of Tumor-Agnostic MRD Detection in Stage III Colorectal Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Feng Wang, Professor, Sun Yat-sen University
Other Study IDs: TRACE-CRC
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer; MRD; ctDNA
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Tissue
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with stage III colorectal cancer
  Interventions: Diagnostic Test: MRD detection

INTERVENTIONS:
Diagnostic Test: MRD detection — Baseline blood samples, surgical resected tumor tissue, blood samples after surgery, and blood samples after adjuvant therapy will be collected from colorectal patients. MRD will be assessed using both tumor-informed and tumor-agnostic methods.

SUMMARY:
This observational study aims to evaluate the predictive performance of various omics-based methods for detecting minimal residual disease (MRD) in stage III colorectal cancer. The study involves the collection of blood samples from patients who have accepted surgery for colorectal cancer. Blood samples will be analyzed using both tumor-informed and tumor-agnostic approaches to detect circulating tumor DNA (ctDNA). The study will compare the sensitivity of these methods and assess their correlation with recurrence risk. The findings aim to inform the development of optimal MRD detection strategies, ultimately providing a robust molecular basis for personalized treatment decisions.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed colorectal cancer.
* Preoperatively assessed as stage III according to the 8th edition UICC/AJCC staging system.
* Deemed eligible for radical resection upon investigator assessment.
* No prior anti-tumor therapy received.
* ECOG PS score 0-1.
* Willing and able to provide signed informed consent for participation in the study.

Exclusion Criteria:

* Has a history of other malignant tumors.
* Pregnant and lactating women.
* Presence of any concurrent medical or psychiatric condition, as assessed by the investigator, that may interfere with protocol compliance, study follow-up, or affect short-term survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 229 patients newly diagnosed with stage III colorectal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 229 (Estimated)
Dates: Start 2025-11-24 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The predictive role of MRD in prognosis | 3 years
  The survival difference between MRD positive and MRD negative patients.

SECONDARY OUTCOMES:
The positive detection rate of baseline ctDNA | 1 year
Predictive Accuracy of MRD for Recurrence | 3 years
  Sensitivity, Specificity, Positive predictive value, and Negative predictive value of ctDNA-MRD in predicting postoperative recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China